CLINICAL TRIAL: NCT04243590
Title: Validity and Reliability of the Turkish Version of Hand-Use-at-Home Questionnaire in Children With Neonatal Brachial Plexus Palsy or Unilateral Cerebral Palsy.
Brief Title: Turkish Version of Hand-Use-at-Home Questionnaire
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 09.2018.712
Record Dates: First submitted 2020-01-24; First posted 2020-01-28 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Palsy; Brachial Plexus Palsy
Keywords: brachial plexus; unilateral cerebral palsy; hand function; child rehabilitation; upper extremity; hand use at home questionnaire
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonatal brachial plexus palsy: 25 patients will be included. The level of the brachial plexus lesion will be recorded. Parents of all patients were asked to fill in the Turkish version of the "Hand-at-Home Questionnaire" and in addition, the upper extremity section of the Pediatric Outcomes Data Collection Instrument (PODCI) in patients with OBP.
  Interventions: Behavioral: Hand-Use-at-Home Questionnaire (HUH); Behavioral: Pediatric Outcome Data Collection Instrument (PODCI)
- Unilateral cerebral palsy: 25 patients will be included. The level of "Manual Ability Classification System (MACS)" will be recorded. Parents of all patients were asked to fill out the Turkish version of the "Hand-at-Home Questionnaire at Home", as well as the "Children's Hand-Use Experience Questionnaire (CHEQ)" in patients with CP.
  Interventions: Behavioral: Hand-Use-at-Home Questionnaire (HUH); Behavioral: Children's Hand-Use Experience Questionnaire (CHEQ)

INTERVENTIONS:
Behavioral: Hand-Use-at-Home Questionnaire (HUH) — The HUH assesses the amount of spontaneous use of the affected hand in children with unilateral upper limb paresis aged 3-10 years, performing 18 typical bimanual play and self-care activities. Parents rate items using a 5-point rating scale (never-sometimes-regularly-often-always). After completion, the ratings are converted into a 3-point score (i.e. never/sometimes = score 0, regularly/ often = score 1, always = score 2). A sum score can be calculated (range 0-36).
Behavioral: Pediatric Outcome Data Collection Instrument (PODCI) — The PODCI is designed to assess different aspects of daily living in children with musculoskeletal disorders. It has excellent psychometric properties, and it is a widely accepted instrument to provide parent/patient-reported information about upper extremity functioning. A Dutch version is available and it is validated for children with neonatal brachial plexus palsy. It consists of 85 questions and five scale scores and one total score can be calculated (range for all scales and total score 0-100, higher scores indicating better functioning/quality of life). Only the Upper Extremity and Physical Function Scale (8 items) were used in this study since this scale provides information about difficulties performing activities using the arms/hands (score 0-100; lower score, more difficulties).
  Groups: Neonatal brachial plexus palsy
Behavioral: Children's Hand-Use Experience Questionnaire (CHEQ) — The CHEQ is a questionnaire for children (aged 6-18) with unilateral functional limitations of hand use and is well validated for children with unilateral cerebral palsy. It was only partially validated for use in children with neonatal brachial plexus palsy and has not yet been used in studies. Therefore, it was not used in this group. The questionnaire consists of 29 bimanual activities, typically requiring the use of both hands. It assesses the child's experience using their affected hand when performing the activities and counts how many of the activities are executed independently (with and without using the affected hand).
  In the mini-version of the CHEQ some items were deleted or replaced (with more age-appropriate activities for children aged three to eight years) and this version was used for all unilateral cerebral palsy children <six years in this study.
  Groups: Unilateral cerebral palsy

SUMMARY:
To investigate the validity and reliability of the Turkish Version of parent-rated Hand-Use-at- Home questionnaire (HUH) in children with neonatal brachial plexus palsy or unilateral cerebral palsy.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is defined as a permanent but non-progressive disorder group that affects the developing fetal or infantile brain, leading to impairment in movement and posture, thereby limiting physical activity and participation. The prevalence of CP in society is around 0.21%. In a study conducted in Turkey, this ratio of 4.4 / 1000 live births has been reported. Motor disorders in CP often are accompanied by sensory, perceptual, cognitive, communicative and behavioral problems and secondary musculoskeletal problems.

Obstetric brachial plexus (OBP) injury is a common peripheral nerve injury in children. Its incidence is reported between 0.42 and 5.1 per 1000 live births. As the primary mechanism of injury, it is accepted that traction or compression of all or part of the brachial plexus.

In these patients, weakness in the upper extremity, long-term contractures, and difficulties in the use of the extremities occurs due to the damage of nerves. In both diseases, patients have difficulty in bimanual activities.

Many treatment methods focus on increasing the use of upper extremities of patients and ensuring their independence in daily life activities. There are many methods for evaluating the hand use performance of patients and the effectiveness of different treatment methods. However, these clinical evaluation methods often do not reflect the patient's performance at home, at school, in their daily living environments.

The "Hand Use at Home (HUH)" questionnaire, which was created to be evaluated by parents, was developed in 2017 for measuring and evaluating the spontaneous use time of unilateral paretic children aged 3-10 in the affected hand and arm daily life activities.

The validity and reliability of the questionnaire were determined in children with obstetric brachial plexus paralysis and unilateral SP.

The purpose of this study; The translation of the HUH questionnaire into Turkish is to investigate its cultural adaptation, validity, and test-retest reliability.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of unilateral cerebral palsy or obstetric brachial plexus palsy
* Age between 3 - 10
* Volunteer to study

Exclusion Criteria:

* Having a visual disorder
* History of botulinum toxin injection and surgery for upper extremity and hand in the last 6 months.
* Having robotic rehabilitation or intensive treatments such as constraint-induced movement therapy to increase upper extremity use in the last 6 months.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 42 unilateral cerebral palsy patients and 25 brachial plexus palsy between 3 - 10 years of age.
Sampling Method: Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-01-24 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Hand-Use-at-Home Questionnaire | Day 0
  The HUH assesses the amount of spontaneous use of the affected hand in children with unilateral upper limb paresis aged 3-10 years, performing 18 typical bimanual play and self-care activities. Parents rate items using a 5-point rating scale (never-sometimes-regularly-often-always). After completion, the ratings are converted into a 3-point score (i.e. never/sometimes = score 0, regularly/often = score 1, always = score 2).
Hand-Use-at-Home Questionnaire (HUH) | Day 7
  The HUH assesses the amount of spontaneous use of the affected hand in children with unilateral upper limb paresis aged 3-10 years, performing 18 typical bimanual play and self-care activities. Parents rate items using a 5-point rating scale (never-sometimes-regularly-often-always). After completion, the ratings are converted into a 3-point score (i.e. never/sometimes = score 0, regularly/often = score 1, always = score 2).

SECONDARY OUTCOMES:
Pediatric Outcome Data Collection Instrument (PODCI) | Day 0
  The PODCI is designed to assess different aspects of daily living in children with musculoskeletal disorders. It has excellent psychometric properties, and it is a widely accepted instrument to provide parent/patient-reported information about upper extremity functioning. It consists of 85 questions and five scale scores and one total score can be calculated (range for all scales and total score 0-100, higher scores indicating better functioning/quality of life). Only the Upper Extremity and Physical Function Scale (8 items) was used in this study since this scale provides information about difficulties performing activities using the arms/hands (score 0-100; lower score, more difficulties).
Children's Hand-Use Experience Questionnaire (CHEQ/mini-CHEQ) | Day 0
  The CHEQ is a questionnaire for children (aged 6-18) with unilateral functional limitations of hand use and is well validated for children with unilateral cerebral palsy. The questionnaire consists of 29 bimanual activities, typically requiring the use of both hands. It assesses the child's experience using their affected hand when performing the activities and counts how many of the activities are executed independently (with and without using the affected hand).
  In the mini-version of the CHEQ some items were deleted or replaced (with more age-appropriate activities for children aged three to eight years) and this version was used for all unilateral cerebral palsy children <six years in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Naime Evrim Karadag Saygi, Prof, Study Director — Department of PM&R, Marmara University School of Medicine; Ayca Evkaya, Res. Asst., Principal Investigator — Department of Physiotherapy and Rehabilitation, Maltepe University; Ayse Simsek, PT (MSc), Principal Investigator — Department of Physiotherapy and Rehabilitation, Gazi University.
Locations (1):
- Marmara University School of Medicine Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Result] Oskoui M, Coutinho F, Dykeman J, Jette N, Pringsheim T. An update on the prevalence of cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2013 Jun;55(6):509-19. doi: 10.1111/dmcn.12080. Epub 2013 Jan 24. PMID 23346889
- [Result] Andersen J, Watt J, Olson J, Van Aerde J. Perinatal brachial plexus palsy. Paediatr Child Health. 2006 Feb;11(2):93-100. doi: 10.1093/pch/11.2.93. PMID 19030261
- [Result] Brandao M, Ocarino JM, Bueno KM, Mancini MC. Hand use at home and in clinical settings by children with cerebral palsy: a qualitative study. Occup Ther Int. 2015 Mar;22(1):43-50. doi: 10.1002/oti.1383. Epub 2014 Oct 29. PMID 25354327
- [Result] van der Holst M, Geerdink Y, Aarts P, Steenbeek D, Pondaag W, Nelissen RG, Geurts AC, Vliet Vlieland TP. Hand-Use-at-Home Questionnaire: validity and reliability in children with neonatal brachial plexus palsy or unilateral cerebral palsy. Clin Rehabil. 2018 Oct;32(10):1363-1373. doi: 10.1177/0269215518775156. Epub 2018 May 13. PMID 29756465